CLINICAL TRIAL: NCT02426840
Title: Effect of Calcium and High-dose Vitamin D Supplementation on Bone Mineral Density Among Perinatally HIV-infected Children and Adolescents
Brief Title: Calcium and High-dose Vitamin D Supplementation on Bone Mineral Density Among HIV-infected Children and Adolescents
Acronym: CAL-D
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Collaborators: HIV-NAT, Thai Red Cross - AIDS Research Centre (Unknown); Nakornping Hospital (Other)
Responsible Party: Principal Investigator, Tavitiya Sudjaritruk, Principle Investigator, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAL-D
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Adverse Bone Health; HIV Infection
Keywords: Adverse bone health; Bone demineralization; HIV-infection; Children; Adolescents; Calcium; Vitamin D; Supplementation
MeSH Terms: conditions — HIV Infections; Bone Demineralization, Pathologic; Acquired Immunodeficiency Syndrome | interventions — Vitamin D; Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High dose vitamin D and calcium (Experimental): Fixed-dose combination (FDC) of 1,500 mg of calcium carbonate (equivalent to 600 mg of elemental calcium) and 200 IU of vitamin D3, administered orally twice daily plus vitamin D2 (20,000 IU/cap) administered once weekly (a total of 1,200 mg of elemental calcium and 3,200 IU of vitamin D daily)
  Interventions: Dietary Supplement: High dose vitamin D and calcium
- Normal dose vitamin D and calcium (Active Comparator): Fixed-dose combination (FDC) of 1,500 mg of calcium carbonate (equivalent to 600 mg of elemental calcium) and 200 IU of vitamin D3, administered orally twice daily (a total of 1,200 mg of elemental calcium and 400 IU of vitamin D daily)
  Interventions: Dietary Supplement: Normal dose vitamin D and calcium

INTERVENTIONS:
Dietary Supplement: High dose vitamin D and calcium — participants will receive a FDC tablet containing 1500 mg of calcium carbonate (equivalent to 600 mg of elemental calcium) and 200 IU of vitamin D3. This drug will be administered as 1 tablet orally twice daily and is to be taken with food. In addition, participants will receive vitamin D2 capsule containing 20,000 IU of ergocalciferol, which will be administered as 1 capsule orally once weekly at any time (not related with meal).
  Arms: High dose vitamin D and calcium
Dietary Supplement: Normal dose vitamin D and calcium — participants will receive a FDC tablet containing 1500 mg of calcium carbonate (equivalent to 600 mg of elemental calcium) and 200 IU of vitamin D3. This drug will be administered as 1 tablet orally twice daily and is to be taken with food
  Arms: Normal dose vitamin D and calcium

SUMMARY:
Since there is no cure for HIV, therefore antiretroviral therapy must be taken life-long. Some of the HIV medications can negatively impact the health of the bone and is even more exacerbated in perinatally HIV-injected children and adolescents because this is the period when the bone peaks. Bone loss during this period can be devastating and increase the risk for developing weak bones later in life. Supplementation of calcium and vitamin D have not been well studied in HIV-infected children and adolescents in developing countries. Therefore it is not clear whether higher doses of these supplementations can thwart the damages or not.

DETAILED DESCRIPTION:
Adverse bone health is one of the major long-term complications among perinatally HIV-infected children and adolescents receiving ART. Since a great deal of bone mineral accrual occurs during the adolescent years and the peak attainment is usually seen at age 18 years, the loss of bone deposition during this period could lead to serious consequences, particularly increased risk of osteoporosis and bone fragility in later of life. A previous study demonstrated that prevalence of low BMD among perinatally HIV-infected Thai children and adolescents was high (25%). However, the prevention strategies such as calcium and vitamin D supplementation which are widely recommended by many guidelines for preventing of osteoporosis and bone fracture have not been well studied to prove their effectiveness among HIV-infected children and adolescents, especially in resource-limited countries. This is considered as the critical research question in pediatric HIV/AIDS field which are urgently required robust and in-depth investigations.

This randomized clinical trial study will provide important information about the effect of calcium and high dose (comparing to normal dose) vitamin D supplementation on BMD among ART-experienced, perinatally acquired HIV-infected children and adolescents to best understand the relative contributions of the supplementation to improve bone health status. This study will address research questions, fill gaps in knowledge, and draw clinician attentions to the important long-term medical complications in children and adolescents who are growing up with HIV. Moreover, this study will inform healthcare providers and policy makers about the importance of calcium and vitamin D supplementation as one of the measurement to prevent long-term deterioration of bone mass and the mean to promote bone health among these populations.

The funding for this study is the National Research University, Chiang Mai University.

ELIGIBILITY:
Inclusion criteria:

* Participants age 10-20 years.
* Have a history and/or medical record of HIV infection.
* Have a history and/or medical record and/or maternal HIV status confirmed of perinatally acquired HIV infection.
* Have virological suppression after receiving ART, defined as plasma HIV RNA less than 400 copies/mL within 12 months prior to screening.
* Participants who had been evaluated for BMD (have BMD result) within 1 year prior to entry visit.
* Caregivers and/or participants gives written inform consent/assent form.

Exclusion criteria:

* Participants who have a documented history of bone fracture at any time prior to screening.
* Participants who have received any form of calcium greater than 1000 mg/day of elemental calcium at least once within 6 months prior screening.
* Participants who have received any form of vitamin D (e.g., ergocalciferol or cholecalciferol) supplementation greater than 400 IU/day at least once within 6 months prior to screening.
* Participants who have received any past pharmacologic treatment for low bone density or osteoporosis (e.g., alendronate) at any time prior to screening.
* Participants who have a documented history of growth hormone deficiency at any time or using growth hormone within 6 months prior to screening.
* Participants who have a documented history of primary hyperparathyroidism, hypoparathyroidism, or cushing syndrome at any time prior to screening.
* Participants who have a documented prior history of kidney stone, renal failure, or renal function impairment (serum creatinine >2 mg/dL).
* Participants who have a documented prior history of chronic active liver diseases, or liver impairment (alanine aminotransferase [ALT] >100 IU/L at least 2 times within 6 months).
* Participants who have a documented prior history of thalassemia major (homozygous β-Thalassemia or β-Thalassemia/Hemoglobin E) or sickle cell disease.
* Participants use any oral, intravenous, or inhaled steroids within 6 months prior to study entry (intranasal steroid use is allowed).
* Participants who have received anticonvulsant medications (phenytoin, phenobarbital, carbamazepine), methotrexate, within 6 months prior to screening.
* Pregnancy or breast feeding
* Participants who have any condition that, in the opinion of the site investigator, would compromise the subject's ability to participate in the study.

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
lumbar spine Bone Mineral Density (BMD) | 48 weeks
  To compare the changes in lumbar spine BMD in perinatally HIV-infected children and adolescents receives 48-week of calcium and high-dose vitamin D supplementation with that of children and adolescents receiving 48-week of calcium and normal dose vitamin D supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Tavitiya Sudjaritruk, MD, Principal Investigator — Chiang Mai University
Locations (5):
- Thailand (5):
  - HIV-NAT, Thai Red Cross - AIDS Research Centre, Bangkok
  - Queen Sirikit National Institute of Child Health, Bangkok
  - Faculty of Medicine and Research Institute for Health Sciences (RIHES), Chiang Mai University, Chiang Mai
  - Nakornping hospital (NKP), Chiang Mai
  - Chiangrai Prachanukroh Hospital, Chiang Rai

REFERENCES:
- [Derived] Sudjaritruk T, Bunupuradah T, Aurpibul L, Kanjanavanit S, Chotecharoentanan T, Sricharoen N, Ounchanum P, Suntarattiwong P, Pornpaisalsakul K, Puthanakit T; CAL-D Study Group. Impact of Vitamin D and Calcium Supplementation on Bone Mineral Density and Bone Metabolism Among Thai Adolescents With Perinatally Acquired Human Immunodeficiency Virus (HIV) Infection: A Randomized Clinical Trial. Clin Infect Dis. 2021 Nov 2;73(9):1555-1564. doi: 10.1093/cid/ciab547. PMID 34125899
- See also: Research Institute for Health Sciences, Chiang Mai University — http://www.rihes.org
- See also: HIV-NAT, Thai Red Cross AIDS Research Center — http://www.hivnat.org